CLINICAL TRIAL: NCT06198543
Title: Study on Exosome Changes in Patients With Proliferative Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: wuhang
Record Dates: First submitted 2023-12-11; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy
Keywords: plasma; aqueous humor; vitreous humor; exosomes; proteomics
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: proliferative diabetic retinopathy
- control group: patients with macular epiretinal membranes and macular holes without diabetes.

SUMMARY:
Diabetic retinopathy is a common complication of diabetes and one of the leading causes of low vision and blindness in adults. In recent years, the prevalence of diabetes and the incidence of diabetic retinopathy have increased significantly in our country. Epidemiological studies show that the prevalence rate of diabetes in China is 12.8%, and the prevalence rate of DR in adult diabetic patients is 24.7%-37.5%, that is, there are about 3200-48 million DR patients in China, and the patients have a trend of younger people. DR has become a serious public health problem threatening people's lives and health.

At present, it is known that the pathogenesis of DR is related to hypoxia, oxidative stress, inflammation, abnormal expression of cytokines and gene methylation, but the specific pathogenesis has not been fully clarified. Due to the hidden early symptoms of DR, the lack of basic screening conditions in primary medical and health institutions, and the lack of awareness of DR by patients themselves, many DR patients have already appeared serious retinopathy when they seek medical treatment, resulting in irreversible visual function impairment. In addition, the current clinical treatment methods for DR mainly include retinal photocoagulation therapy, intraocular anti-VEGF drug injection and vitrectomy surgery, etc. These methods are aimed at relatively severe diabetic retinopathy, and there is no effective treatment method for early diabetic retinopathy that can prevent or slow down the occurrence and development of DR. Therefore, to further explore the pathogenesis of DR and develop new therapeutic methods has become an urgent problem.

Exosomes are extracellular vesicles secreted by living cells with a diameter of 40-150nm. With a bilayer lipid membrane structure, exosomes contain a variety of biomolecules such as lipids, proteins, nucleic acids, cytokines, and autoantigens, and are important mediators for the transmission of biological information between cells. Almost all cells can secrete exosomes, and exosomes from different cells have different functions. Exosomes transfer their contents to nearby or distant cells and participate in cell growth, angiogenesis, immune regulation and other processes. Previous studies have shown that exosomes secreted by various cells in the retina are present in the vitreous and aqueous humor of patients and play an important role in the pathogenesis of DR. At the same time, exosomes in the systemic circulation of diabetic patients can also reach the retina through the blood circulation, participate in the initiation process of DR And play an important role. At the same time, due to the double-layer lipid membrane structure, exosomes can also target the coated components to specific cells and tissues through biological barriers such as blood-brain and blood-eye, which is expected to become a highly efficient drug delivery route. Therefore, the role of exosomes in DR Treatment has also attracted much attention.

DETAILED DESCRIPTION:
一、Research Purpose

1. compared the changes of exosomes in intraocular fluid and blood of patients with proliferative diabetic retinopathy and non-diabetic patients.
2. analysed differentially expressed proteins in the exosomes of the two groups of patients using proteomic techniques, laying the foundation for screening possible biomarkers and potential therapeutic targets for the early diagnosis of diabetic retinopathy.

二、Design

1. Subject Population Patients with proliferative diabetic retinopathy and non-diabetic macular epiretinal membrane/macular hole requiring vitrectomy were admitted to the Ophthalmology Department of Xuanwu Hospital, Capital Medical University.
2. Sample Size A total of 60 patients were included in the study.
3. Grouping of Subjects Experimental group: proliferative diabetic retinopathy; Control group: patients with macular epiretinal membranes and macular holes without diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Patients diagnosed with PDR by FFA and requiring vitrectomy for treatment;
3. Patients with no history of diabetes and diagnosed with macular anterior membrane or macular hiatus by color fundus photography and OCT;
4. Sign the informed consent form.

Exclusion Criteria:

1. Suffering from cancer, immune diseases, infectious diseases and other systemic diseases;
2. Patients with retinal arteriovenous obstruction;
3. Intraocular infection;
4. Patients with uveitis;
5. In patients with high myopia, the equivalent spherical lens was > -9.0D;
6. Recent history of cerebral infarction, myocardial infarction and other thrombus;
7. Patients with contraindications to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects enrolled in this study were patients over 18 years of age who signed an informed consent form requiring vitrectomy treatment. Subjects in the experimental group were patients with proliferative diabetic retinopathy, and those in the control group were patients who did not have diabetes but had macular holes or epiretinal membranes. Those with the following conditions could not be enrolled in the study:1) Suffering from cancer, immune diseases, infectious diseases and other systemic diseases;2) Patients with retinal arteriovenous obstruction;3) Intraocular infection;4) Patients with uveitis;5) In patients with high myopia, the equivalent spherical lens was > -9.0D;6) Recent history of cerebral infarction, myocardial infarction and other thrombus;7) Patients with contraindications to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
differential proteins of exosomes | January 2024 - January 2025
  Exosomes from plasma, atrial fluid and vitreous fluid were isolated and extracted, and proteomic analysis of proteins in exosomes was performed to analyse the number of differentially expressed protein species in the test and control groups, and bioinformatics analysis of up-regulated or down-regulated expressed proteins was performed.